CLINICAL TRIAL: NCT05890235
Title: Efficacy and Safety of Ningmitai Capsule in Patients With Chronic Prostatitis/Chronic Pelvic Pain Syndrome：A Prospective, Randomized, Positive Drug-controlled, Multicenter Clinical Study
Brief Title: Efficacy and Safety of Ningmitai Capsule in Patients With Chronic Prostatitis/Chronic Pelvic Pain Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xintian Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMT18016S
Record Dates: First submitted 2023-05-23; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Chronic Prostatitis
MeSH Terms: interventions — Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ningmitai Capsule group (Experimental): Patients take Ningmitai capsule, 0.38 g/capsule, tid, 4 capsules each time, after meals, for 8 weeks.
  Interventions: Drug: Ningmitai Capsule
- Tamsulosin Hydrochloride Sustained-release Capsules group (Active Comparator): Patients take Tamsulosin Hydrochloride Sustained-release Capsules ,0.2 mg/capsule, once daily, 1 capsule each time, for 8 weeks.
  Interventions: Drug: Tamsulosin Hydrochloride
- Combined group (Active Comparator): Patients take Ningmitai capsule, 0.38 g/capsule, tid, 4 capsules each time, after meals, for 8 weeks and Tamsulosin Hydrochloride Sustained-release Capsules ,0.2 mg/capsule, once daily, 1 capsule each time, for 8 weeks.
  Interventions: Drug: Ningmitai Capsule; Drug: Tamsulosin Hydrochloride

INTERVENTIONS:
Drug: Ningmitai Capsule — Ningmitai Capsule (Ningmitai®) is Traditional Chinese Medicine which has already used in treatment of urinary system disease (eg. CPPS, BPH) in China for more than twenty years. The instruction of Ningmitai Capsule is 0.38g/capsule, 4 capsule/time, tid.
  Other Names: Ningmitai
  Arms: Combined group; Ningmitai Capsule group
Drug: Tamsulosin Hydrochloride — Tamsulosin is α1A-adrenergic receptor which has used in treatment of BPH for few years. The instruction of Tamsulosin Capsule is 1 tablet at a time, 1 time a day.
  Other Names: Tamsulosin
  Arms: Combined group; Tamsulosin Hydrochloride Sustained-release Capsules group

SUMMARY:
1. Clinical trial title：Efficacy and safety of Ningmitai capsule in patients with Chronic Prostatitis/Chronic Pelvic Pain Syndrome：A prospective, randomized, positive drug-controlled, multicenter clinical study
2. Version number/date：1.0 /2018-6-24
3. Principal investigator：Zhang Xiansheng
4. Main research units：The first affiliated hospital of Anhui medical university clinical medical research ethics committee
5. Clinical trial start and end dates：2018-10-1-2022-12-31
6. Objective: To observe whether Ningmitai capsule(NMT) alone or combined with Tamsulosin for 8 weeks is more effective than Tamsulosin in improving symptoms of CP/CPPS .
7. Study type:Interventional study
8. Total sample size:300
9. Inclusion criteria:

   ① Age: male patients aged 18-60 years;

   ② Long-term and repeated pelvic discomfort or pain (NIH-CPSI pain score ≥ 4 points), lasting more than 3 months, may be accompanied by different degrees of urination symptoms and sexual dysfunction;

   ③ Diagnosed as type III prostatitis.

   Exclusion criteria:
   * Use any antibiotics and α1 receptor blockers in the past two weeks; ② Suffering from seminal vesiculitis, epididymitis, varicocele, tumors in prostate, bladder and urethra and other diseases affecting bladder function;

     * Have received transurethral resection of the prostate(TURP), transurethral incision of the prostate (TUIP), bladder neck incision, transurethral hyperthermia/radiofrequency ablation/balloon dilatation, open prostatectomy, or any other prostate surgery and treatment, such as cryotherapy;

       * Patients with severe cardiovascular and cerebrovascular diseases, liver, kidney and hematopoietic diseases and psychosis; ⑤ Patients who are allergic to NMT or some of its components; ⑥ Patients who are involuntarily unable to cooperate with the completion of the test.
10. Interventions:

1. NMT group Oral Ningmitai capsule, 0.38 g/capsule, tid, 4 capsules each time, after meals, for 8 weeks.

Sample size:100 2. Tamsulosin group Tamsulosin Hydrochloride Sustained-release Capsules were orally administered at 0.2 mg/capsule, once daily, 1 capsule each time, for 8 weeks.

Sample size:100 3.Combination group Oral Ningmitai capsule, 0.38 g/capsule, tid, 4 capsules each time, after meals, for 8 weeks.Tamsulosin Hydrochloride Sustained-release Capsules were orally administered at 0.2 mg/capsule, once daily, 1 capsule each time, for 8 weeks.

Sample size:100

DETAILED DESCRIPTION:
1. Clinical trial title：Efficacy and safety of Ningmitai capsule in patients with Chronic Prostatitis/Chronic Pelvic Pain Syndrome：A prospective, randomized, positive drug-controlled, multicenter clinical study
2. Version number/date：1.0 /2018-6-24
3. Principal investigator：Zhang Xiansheng
4. Main research units：The first affiliated hospital of Anhui medical university clinical medical research ethics committee
5. Clinical trial start and end dates：2018-10-1-2022-12-31
6. Objective: To observe whether Ningmitai capsule(NMT) alone or combined with Tamsulosin for 8 weeks is more effective than Tamsulosin in improving symptoms of CP/CPPS .
7. Study type:Interventional study
8. Total sample size:300
9. Interventions:

1. NMT group Oral Ningmitai capsule, 0.38 g/capsule, tid, 4 capsules each time, after meals, for 8 weeks.

Sample size:100 2. Tamsulosin group Tamsulosin Hydrochloride Sustained-release Capsules were orally administered at 0.2 mg/capsule, once daily, 1 capsule each time, for 8 weeks.

Sample size:100 3.Combination group Oral Ningmitai capsule, 0.38 g/capsule, tid, 4 capsules each time, after meals, for 8 weeks.Tamsulosin Hydrochloride Sustained-release Capsules were orally administered at 0.2 mg/capsule, once daily, 1 capsule each time, for 8 weeks.

Sample size:100

10、Treatment cycle：8 weeks. the trial treatment began on the day of randomization.

11、Visiting nodes：① before treatment (-2 weeks to 0 days), ②4 weeks of treatment (28 ± 10 days), ③ 8 weeks of treatment (56 ± 14 days).

12、Countries of recruitment and research settings: Country:China Province:Anhui Institution(hospital):The first affiliated hospital of Anhui medical university Level of the institution:Tertiary A

13、Recruiting status:Completed Participant age:18 years Participant age:60 years Gender: Male

14、Randomization Procedure:In this study, the research center was used as the stratification factoror random assignment. Subjects were randomly assigned (1:1:1) to Tamsulosin group, NMT group and combination group according to the random allocation table (subject random code) simulated by SAS 9.2 software. Subjects' random numbers cannot be reused by other subjects, whether they are using the study drug or not, or the study is terminated for any reason.

15、Sign the informed consent: Yes

16、Data collection and Management (A standard data collection and management system include a CRF and an electronic data capture:In this study, case report form (CRF) was used to collect and manage research data. The sponsor or designated person is responsible for data management of the study, including data quality control. The workflow of data management includes data entry, data verification and query, medical coding, data audit, database locking, data export and transmission, data and data management file archiving, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-60 years old male patients;
2. Patients with long-term, repeated pelvic discomfort or pain (NIH-CPSI pain score 4), lasting more than 3 months, may be accompanied by varying degrees of voiding symptoms and sexual dysfunction.
3. Clinical diagnosis: type III prostatitis.

Exclusion Criteria:

1. Use of any antibiotics and 1 receptor blockers in the past two weeks;
2. Suffering from seminal vesiculitis, epididymitis, varicocele and prostate, bladder, urethra and other tumors and other diseases affecting bladder function;
3. Have received TURP, TUIP, internal cystotomy, transurethral hyperthermia/radiofrequency ablation/balloon dilatation, open prostatectomy, or any other prostate surgery and treatment, such as cryotherapy or hyperthermia;
4. Patients with severe cardiovascular and cerebrovascular, liver, kidney and hematopoietic system diseases and mental illness;
5. Known to be allergic to Ningmitai capsule or some of its components;
6. Involuntary, unable to cooperate with the completion of the study.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 323 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
The National Institutes of Health chronic prostatitis symptom index total score | Treatment for 8 weeks
  the change of NIH-CPSI total score from baseline to 8 weeks. National Institutions of Health Chronic Prostatitis Symptom Index（NIH-CPSI，0~43 points） consists of three subscales. The first part is pain symptoms, which consists of questions 1~4 (0~21 points), and evaluates the location, frequency and severity of pain. The second part is urination symptoms, which consists of questions 5~6 (0 ~ 10 points), and evaluates the severity of incomplete urination and frequent urination; The third part is to evaluate the impact on the quality of life, which consists of questions 7~9 (0~12 points).The higher the score, the more serious the symptoms of chronic prostatitis.

SECONDARY OUTCOMES:
NIH-CPSI total score, pain score, urinary score and quality of life score | Treatment for 4 weeks
  The changes of NIH-CPSI total score, pain score, urinary score and quality of life score from baseline to 4 weeks; National Institutions of Health Chronic Prostatitis Symptom Index（NIH-CPSI，0~43 points） consists of three subscales. The first part is pain symptoms, which consists of questions 1~4 (0~21 points), and evaluates the location, frequency and severity of pain. The second part is urination symptoms, which consists of questions 5~6 (0 ~ 10 points), and evaluates the severity of incomplete urination and frequent urination; The third part is to evaluate the impact on the quality of life, which consists of questions 7~9 (0~12 points).The higher the score, the more serious the symptoms of chronic prostatitis.
NIH-CPSI total score, pain score, urinary score and quality of life score | Treatment for 8 weeks
  The changes of NIH-CPSI pain score, urinary score and quality of life score from baseline to 8 weeks; National Institutions of Health Chronic Prostatitis Symptom Index（NIH-CPSI，0~43 points） consists of three subscales. The first part is pain symptoms, which consists of questions 1~4 (0~21 points), and evaluates the location, frequency and severity of pain. The second part is urination symptoms, which consists of questions 5~6 (0 ~ 10 points), and evaluates the severity of incomplete urination and frequent urination; The third part is to evaluate the impact on the quality of life, which consists of questions 7~9 (0~12 points).The higher the score, the more serious the symptoms of chronic prostatitis.
Response rate | Treatment for 4 & 8 weeks
  The response rate is defined as a decrease of at least 25% in the NIH-CPSI total score and pain score, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Zhongguo Chen, MD, Study Chair — employee
Locations (1):
- The first affiliated hospital of Anhui medical university, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao J, Zhang Y, Du J, Liu Q, Cheng Y, Yang W, Wang D, Wang W, Zheng L, Wang D, Wu L, Jiang X, Men Q, Liang C, Zhang X. Ningmitai capsule in patients with chronic prostatitis/chronic pelvic pain syndrome: a multicenter, prospective, randomized, parallel, positive-controlled study. Front Pharmacol. 2025 Dec 3;16:1667819. doi: 10.3389/fphar.2025.1667819. eCollection 2025. PMID 41415574